CLINICAL TRIAL: NCT00001067
Title: A Phase II Randomized Study of the Virologic and Immunologic Effects of Zidovudine Plus Lamivudine (3TC) Versus d4T Versus Zidovudine Plus d4T in HIV-Infected Patients With CD4 Cell Counts Between 300-600/mm3 and No Previous Nucleoside Experience
Brief Title: The Effectiveness of Three Anti-HIV Drug Combinations in HIV-Infected Patients Who Have Never Used Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 298; 11274 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; Stavudine; Lamivudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To determine drug efficacy and safety in HIV-infected patients treated with zidovudine ( AZT ) versus stavudine ( d4T ) versus both drugs. Also, to compare short- and long-term changes in magnitude of HIV RNA over time.

Asymptomatic patients with CD4 counts over 300 cells/mm3 are more likely to tolerate any of the nucleoside analogs. d4T, with a favorable toxicity profile and demonstrated anti-HIV activity in previous studies, provides an additional therapeutic option.

DETAILED DESCRIPTION:
Asymptomatic patients with CD4 counts over 300 cells/mm3 are more likely to tolerate any of the nucleoside analogs. d4T, with a favorable toxicity profile and demonstrated anti-HIV activity in previous studies, provides an additional therapeutic option.

Patients are randomized to receive d4T alone, AZT alone, or both in combination for at least 12 weeks. After week 12, 3TC is added to the combination arm. Treatment continues for up to 48 weeks (was a total of 48 weeks, amended 3/26/96).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* TMP / SMX, aerosolized pentamidine, or dapsone for PCP prophylaxis.

Allowed:

* Atovaquone.
* IV pentamidine.
* TMP / SMX.
* Trimetrexate.
* Trimethoprim-dapsone.
* Clindamycin-primaquine.
* Topical antifungals.
* Clotrimazole.
* Ketoconazole.
* Fluconazole.
* Amphotericin B.
* Itraconazole.
* Rifabutin.
* Isoniazid.
* Pyrazinamide.
* Clofazimine.
* Clarithromycin.
* Azithromycin.
* Ethambutol.
* Amikacin.
* Ciprofloxacin.
* Ofloxacin.
* Pyrimethamine.
* Sulfadiazine.
* Clindamycin.
* Filgrastim ( G-CSF ).
* Up to 1000 mg/day acyclovir.
* Erythropoietin.
* Antibiotics.
* Antipyretics.
* Analgesics.
* Antiemetics.
* Rifampin.

Concurrent Treatment:

Allowed:

* Local radiation therapy.

Patients must have:

* HIV infection.
* CD4 count 300 - 600 cells/mm3.
* NO history of AIDS.
* NO active opportunistic infection.
* NO prior nucleoside therapy.
* Life expectancy at least 2 years.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Serious underlying medical condition other than HIV such that life expectancy is less than 2 years.
* Malignancy requiring systemic cytotoxic chemotherapy.
* Active grade 2 or worse peripheral neuropathy.

Concurrent Medication:

Excluded:

* Antiretrovirals other than study drugs.
* Systemic cytotoxic chemotherapy.
* Foscarnet.

Patients with the following prior conditions are excluded:

* Chronic diarrhea defined as three or more stools per day for 15 days, within 30 days prior to study entry.
* Unexplained temperature >= 38.5 C for any 7 days within 30 days prior to study entry.
* Active participation in other experimental therapy within 30 days prior to study entry.

Prior Medication:

Excluded:

* Prior nucleoside antiretrovirals of 1 week or longer duration.
* Any antiretroviral within 90 days prior to study entry.
* Non-nucleoside reverse transcriptase inhibitors and protease inhibitors within 30 days prior to study entry.
* Biologic response modifiers such as IL-2 and interferon within 30 days prior to study entry.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105
Dates: Study Completion 1997-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Havlir D, Study Chair; Pollard R, Study Chair; Richman D, Study Chair; Friedland G, Study Chair
Locations (13):
- United States (12):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Cadman J. 2, 4, 6, 8, who's afraid to phosphorylate? GMHC Treat Issues. 1998 Feb;12(2):6-8. PMID 11365218
- [Background] Havlir DV, Friedland G, Pollard R, Tierney C, Smeaton L, Fox L, Richman DD. Combination zidovudine (ZDV) and stavudine (d4T) therapy versus other nucleosides: report of two randomized trials (ACTG 290 and 298). Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:79 (abstract no 2)
- [Background] Pollard RB, Tierney C, Havlir D, Tebas P, Fox L, Smeaton L, Richman D, Friedland GH. A phase II randomized study of the virologic and immunologic effect of zidovudine + stavudine versus stavudine alone and zidovudine + lamivudine in patients with >300 CD4 cells who were antiretroviral naive (ACTG 298). AIDS Res Hum Retroviruses. 2002 Jul 1;18(10):699-704. doi: 10.1089/088922202760072311. PMID 12167276